CLINICAL TRIAL: NCT03997617
Title: Pilot Study to Explore the Integrated Personalized Functional Profiling (PFP) for Cancer Patients With Metastatic Gastrointestinal Cancer (mGIC) or Recurrent Glioblastoma (rGBM) in Luxembourg
Brief Title: Personalized Functional Profiling in Metastatic Gastrointestinal Cancer or Recurrent Glioblastoma Patients in Luxembourg.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Integrated Biobank of Luxembourg (Other); Laboratoire National de Santé (Luxembourg) (Unknown); Centre Hospitalier du Luxembourg (Other); Hopitaux Robert Schuman (Luxembourg) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PFP-001
Record Dates: First submitted 2019-03-11; First posted 2019-06-25 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized Functional Profiling (Other)
  Interventions: Diagnostic Test: Personalized Functional Profiling

INTERVENTIONS:
Diagnostic Test: Personalized Functional Profiling — During this pilot study, the overall goal of the project is to establish an effective workflow between the patient, the PFP platform, the clinician and return to the patient. This includes collection of the biopsy or surgery piece and standardized processing, dissociation, drug profiling and issuing treatment recommendation to the clinician. In case the clinician follows this treatment recommendation, patient management and follow up will be performed according to standard of care.

SUMMARY:
The investigators are developing a novel standardized and centralized approach named Integrated Personalized Functional Profiling (PFP) in Luxembourg. Based on recent improvements in cancer biopsy-derived 3D-culture technologies the PFP process will screen patient derived cells (PDCs) with FDA/EMA-approved drugs to generate personalized functional response profiles. The selected drug through PFP technology will provide personalized treatment recommendation for the patient.

This pilot study will evaluate the clinical feasibility of setting-up an effective workflow as a first step. Outcomes from this study will be used subsequently to help plan the clinical validation of the implementation of PFP.

ELIGIBILITY:
Inclusion Criteria:

* Patient with recurrent Glioblastoma (rGBM) or with metastatic gastrointestinal cancer (mGIC), i.e. adenocarcinoma (any grade) of stomach, liver, pancreas, small intestine, colon, rectum
* The patient has received previous cancer treatment for mGIC or rGBM
* Male or female ≥ 18 years
* Life expectancy ≥ 12 weeks
* Histologically or cytologically confirmed diagnosis for mGIC or recurrence of a glioblastoma, WHO grade IV
* For women of childbearing potential, a negative pregnancy test documented prior to the screening visit is required
* Signed Inform Consent Form before any study related procedure

Exclusion Criteria:

* For female patient, being pregnant, planning a pregnancy or breastfeeding
* No fresh and viable tumor material available
* Known active Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection
* Uncontrolled medical conditions (i.e, diabetes mellitus, hypertension, etc), psychological, familial, sociological, or geographical conditions that do not allow compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol
* In mGIC arm, patient with non-adenocarcinoma gastrointestinal cancer
* Patient unable to understand and consent himself

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients for which a treatment recommendation for their specific cancer can be formulated, based on PFP | 4 weeks

SECONDARY OUTCOMES:
Quantity of cells needed for the PFP analysis | 4 weeks
Duration of the PFP process for one specific patient | 4 weeks
Number of drugs recommended by using the PFP approach | 4 weeks
Number of patients for which the treatment recommendation issued by PFP were followed by the investigator | 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Luxembourg (2):
  - Centre hospitalier de Luxembourg, Luxembourg, Luxembourg
  - Hôpitaux Robert Schmuan, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No